CLINICAL TRIAL: NCT01374646
Title: Effects of a Community-based Program to Treat Childhood and Adolescent Obesity
Brief Title: Community-based Program to Treat Childhood Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UnitedHealth Group (Industry)
Responsible Party: Dr. Deneen Vojta, UnitedHealth Group
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JOIN2011 10-309
Record Dates: First submitted 2011-06-14; First posted 2011-06-16 (Estimated); Last update posted 2021-06-23 (Actual); Status verified 2021-06

CONDITIONS: Childhood Obesity
Keywords: Childhood Obesity; Group Treatment; Community-based Programs
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: JOIN Intervention — Behavioral group treatment for overweight and obese children and teens, that focuses on decreasing energy dense foods and sedentary behaviors.

SUMMARY:
This study will evaluate the effectiveness of a comprehensive community based program on reducing excess weight in children and teens. This study will recruit 150 participants between the ages of 6-12 and 13-17.

DETAILED DESCRIPTION:
This study will evaluate the effectiveness of a comprehensive community based program on reducing excess weight. Overweight and obese study participants will be grouped with peers of similar ages and their parent/guardians. The participants will be divided into 2 groups, child (6-12 yrs. old) and teens (13-17 yrs. old) and will be accompanied by their parent/guardian. 150 participants will be recruited for this study.

This 6-month program (12 in-person group workshop sessions and 12 at-home sessions) takes the best components of current evidence for individual treatment and places them in a comprehensive community based program. These include:

* Parental involvement
* Reduction in consumption of sugar sweetened beverages
* Reduction of screen time
* Self-monitoring
* Physical activity
* Stimulus control

ELIGIBILITY:
Inclusion Criteria

* Children and teens between the ages of 6-17
* BMI percentile ≥85
* Participation of a parent/guardian

Exclusion Criteria:

* Enrollment in another weight loss program or study
* Diagnosis of type 1 or type 2 diabetes
* Pre-existing medical conditions (e.g., Prader Willi) that affect weight and appetite
* Medications (e.g., steroids) that affect weight or appetite
* Serious or unstable medical or psychological conditions that, in the opinion of the Principal Investigator, would compromise the participant's safety or successful participation in the study

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 155 (Actual)
Dates: Start 2011-01-01 (Actual); Primary Completion 2012-06-05 (Actual); Study Completion 2012-06-05 (Actual)

PRIMARY OUTCOMES:
Change in weight and body mass index (BMI) in children and teens at 6 months | 6 Months
  Assess the effects of a community based program on weight change in children ages 6-12 and teens ages 13-17. Assessments will occur at baseline, 3 and 6 months.

SECONDARY OUTCOMES:
Change in weight and BMI in parent/guardian/care giver at 6 months | 6 months
  Assess the effects of a community based program on weight change in parent/guardian/care givers. Assessments will occur at baseline, 3 and 6 months.
Change in physical activity level in children and teens at 6 months | 6 months
  Assess the effects of a community based program on physical activity level. Accelerometers will be used to access change at baseline, 3 and 6 months.
Changes in intake and sedentary behavior at 6 months | 6 months
  Change in the number of sugar sweetened beverages consumed per day, hours per day on screen time (TV, video games, and computer), and quality of life at 6 months. Assessments will occur at baseline, 3 and 6 months.
Process Outcomes | 6 Months
  Assess process outcomes measures, such as attendance and program satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Deneen Votja, MD, Principal Investigator — UnitedHealth Group
Locations (1):
- YMCA of Greater Providence, Providence, Rhode Island, United States